CLINICAL TRIAL: NCT02491476
Title: Feasibility and Interest of Recording "Fast Ripples" Using Microelectrodes During Stereo-encephalography in Patients With Drug-resistant Partial Epilepsy
Brief Title: Recording "Fast Ripples" Using Microelectrodes During Stereo-encephalography in Patients With Drug-resistant Partial Epilepsy
Acronym: Epi-FaR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: CerCo, CNRS Cerco UMR5549 CHU Purpan Toulouse France (Unknown); DIXI Medical, Besançon, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/13/6899; 2014-A00747-40 (Other: ID-RCB)
Record Dates: First submitted 2015-06-01; First posted 2015-07-08 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2023-06

CONDITIONS: Epilepsy
Keywords: Safety; Electrodes; Device; StereoElectroencephalograph; Epileptogenic zone; Fast ripples
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- micro-macroelectrodes (Experimental): All patients will be implanted with usually 4 intracerebral micro-macroelectrodes(replacing the regular clinical macroelectrodes). The primary and secondary outcomes will then be assessed.
  Interventions: Device: intracerebral micro-macroelectrodes

INTERVENTIONS:
Device: intracerebral micro-macroelectrodes — All patients will be implanted with usually 4 micro-macroelectrodes (replacing the regular clinical macroelectrodes). The primary and secondary outcomes will then be assessed.

SUMMARY:
The main objective of this study is to evaluate the feasibility of recording fast-ripples, a potential new biomarker of epilepsy, using the new micro-macroelectrodes developed by Dixi-Medical.

DETAILED DESCRIPTION:
Partial epilepsies are refractory to medical treatment in 30% of the cases (Refractory Partial Epilepsy or RPE). Patients with RPE suffer from social and occupational disability, an increased risk associated with seizures (traumatic brain injury, accidents), but also a higher risk of sudden unexplained death (2 to 3 times higher) than the general population. Moreover, the medical and social burden of these patients is heavy, representing a significant cost to society.

In some cases, surgical treatment with resection of the epileptogenic zone (EZ) can be proposed. The presurgical evaluation includes various investigations seeking to clarify the location of the EZ; but this approach is sometimes insufficient and the definition of the EZ then requires invasive exploration through intracerebral EEG recording (stereo-EEG, SEEG). This latter technique is currently the preferred standard to define the EZ. It involves implanting electrodes in the brain areas suspected to belong to the seizure network. 50 to 70% of patients investigated with this technique will have epilepsy surgery.

In recent years, a series of studies in animals and humans have suggested that some oscillations, very short and at very high frequency (> 250 Hz), called "fast ripples" (FRs) could be a good biomarker of the EZ (for a review see Zijlmans et al, 2012). The FRs are more easily recorded from microelectrode (diameter: 20-40 microns).

The purpose of this study is to evaluate a new medical device designed by DixiMedical to record FRs, combining micro and regular clinical electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with RPE in whom SEEG is required to precisely localize the seizure focus

Exclusion Criteria:

Patients with SEEG contra-indication:

* severe psychiatric disorders,
* severe agitation during their crisis
* contraindication for performing an MRI: claustrophobia, a cardiac or neural stimulator, ferromagnetic surgical clips, cochlear implants, intraocular metallic foreign body or in the nervous system,
* contraindication to intracerebral investigation (macro-electrodes): ongoing infection, severe associated pathology (cardiac, pulmonary, renal, hepatic), pregnant or nursing women,
* anti thrombotic ongoing treatment.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of the feasibility of recording Fast Ripples (FRs) | During 5 days
  Proportion of patients who are registered more than 60 FRs per hour the day 3 and the day 4 on the micro-macro electrode in the presumed epileptogenic zone, compared to the number of patients included

SECONDARY OUTCOMES:
Evaluation of the interest of FRs | During 5 days
  Sum of FRs recorded over the 5 days.
Evolution of the hourly frequency of FRs | During 5 days
  The evolution of the hourly frequency of FRs recorded by the microelectrodes depending on the day of recording.
Effectiveness of microelectrodes and macroelectrodes | During 5 days
  Number of FRs stored on the macro-blocks immediately adjacent to the microelectrodes located in the EZ.
safety of micro-macroelectrodes | During 5 days
  A quantitative and qualitative description of the side effects associated with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: luc valton, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, Midi-Pyrenees, France

REFERENCES:
- [Background] Bragin A, Wilson CL, Staba RJ, Reddick M, Fried I, Engel J Jr. Interictal high-frequency oscillations (80-500 Hz) in the human epileptic brain: entorhinal cortex. Ann Neurol. 2002 Oct;52(4):407-15. doi: 10.1002/ana.10291. PMID 12325068
- [Background] Crepon B, Navarro V, Hasboun D, Clemenceau S, Martinerie J, Baulac M, Adam C, Le Van Quyen M. Mapping interictal oscillations greater than 200 Hz recorded with intracranial macroelectrodes in human epilepsy. Brain. 2010 Jan;133(Pt 1):33-45. doi: 10.1093/brain/awp277. Epub 2009 Nov 17. PMID 19920064
- [Background] Demont-Guignard S, Benquet P, Gerber U, Biraben A, Martin B, Wendling F. Distinct hyperexcitability mechanisms underlie fast ripples and epileptic spikes. Ann Neurol. 2012 Mar;71(3):342-52. doi: 10.1002/ana.22610. PMID 22451202
- [Background] Jacobs J, Levan P, Chatillon CE, Olivier A, Dubeau F, Gotman J. High frequency oscillations in intracranial EEGs mark epileptogenicity rather than lesion type. Brain. 2009 Apr;132(Pt 4):1022-37. doi: 10.1093/brain/awn351. Epub 2009 Mar 18. PMID 19297507
- [Background] Jacobs J, Zijlmans M, Zelmann R, Chatillon CE, Hall J, Olivier A, Dubeau F, Gotman J. High-frequency electroencephalographic oscillations correlate with outcome of epilepsy surgery. Ann Neurol. 2010 Feb;67(2):209-20. doi: 10.1002/ana.21847. PMID 20225281
- [Background] Staba RJ, Frighetto L, Behnke EJ, Mathern GW, Fields T, Bragin A, Ogren J, Fried I, Wilson CL, Engel J Jr. Increased fast ripple to ripple ratios correlate with reduced hippocampal volumes and neuron loss in temporal lobe epilepsy patients. Epilepsia. 2007 Nov;48(11):2130-8. doi: 10.1111/j.1528-1167.2007.01225.x. Epub 2007 Jul 28. PMID 17662059
- [Background] Worrell GA, Gardner AB, Stead SM, Hu S, Goerss S, Cascino GJ, Meyer FB, Marsh R, Litt B. High-frequency oscillations in human temporal lobe: simultaneous microwire and clinical macroelectrode recordings. Brain. 2008 Apr;131(Pt 4):928-37. doi: 10.1093/brain/awn006. Epub 2008 Feb 7. PMID 18263625
- [Background] Zijlmans M, Jiruska P, Zelmann R, Leijten FS, Jefferys JG, Gotman J. High-frequency oscillations as a new biomarker in epilepsy. Ann Neurol. 2012 Feb;71(2):169-78. doi: 10.1002/ana.22548. PMID 22367988
- [Result] Despouy E, Curot J, Denuelle M, Deudon M, Sol JC, Lotterie JA, Reddy L, Nowak LG, Pariente J, Thorpe SJ, Valton L, Barbeau EJ. Neuronal spiking activity highlights a gradient of epileptogenicity in human tuberous sclerosis lesions. Clin Neurophysiol. 2019 Apr;130(4):537-547. doi: 10.1016/j.clinph.2018.12.013. Epub 2019 Jan 30. PMID 30785010